CLINICAL TRIAL: NCT00834509
Title: Towards a Blood Test for Diagnosis of Obstructive Sleep Apnea
Brief Title: Biomarkers for Obstructive Sleep Apnea
Acronym: BOSA
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Allan Pack, Principal Investigator, University of Pennsylvania
Other Study IDs: 807416; P01HL094307 (NIH)
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary outcome variables: tumor necrosis factor alpha (TNFα); plasma norepinephrine, and free fatty acids. Secondary biomarkers: Interleukin 6 (IL-6), urinary norepinephrine; urinary normetanephrine; glucose, Intercellular Adhesion Molecule (ICAM), leptin. Monocytes will be separated from each blood sample (before, during and after sleep) and RNA extracted. Expression of key genes will be assessed by RT-PCR and microarray studies will be performed in a subset of subjects to assess changes in expression of all genes as a result of OSA. We will evaluate: a)whether individuals with comorbidities have more oxidative stress and inflammatory change for equivalent degrees of OSA than individuals without such comorbidities; b) whether individuals with comorbidities have lower levels of protective mechanisms-melatonin, IL-10; c) different gene variants based on a genetic association study using a recently developed CV SNP array.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea (OSA): OSA participants will be treated with a CPAP/APAP treatment, per standard clinical care.
  Interventions: Device: CPAP
- Control: Control participants will not receive APAP/CPAP treatment, if not diagnosed with OSA.

INTERVENTIONS:
Device: CPAP — Use CPAP for 4-6 weeks as clinically prescribed.
  Groups: Obstructive Sleep Apnea (OSA)

SUMMARY:
The purpose of the study is to:

* recruit subjects with untreated sleep apnea; assess overnight changes in their blood and urine chemicals
* review the overnight changes in blood and urine chemicals after they have been treated for sleep apnea
* assess the overnight changes in blood and urine chemicals in healthy individuals with no sleep problems
* compare the amount of fat in the belly using a Magnetic Resonance Imaging (MRI) scanner on all subjects

DETAILED DESCRIPTION:
The overall goal of this project is to address the postulate that the optimal molecular signature for the common disorder obstructive sleep apnea (OSA) is change in relevant biomarkers during the sleep period. In sleep apnea, events lead to sleep fragmentation and cyclical deoxygenation/reoxygenation. It is proposed that these changes will lead to molecular consequences can be detected by assessing biomarkers in blood. To determine which changes are due to OSA and which to circadian/sleep mechanisms, studies will be done in patients with OSA before and after effective treatment with Continuous Positive Airway Pressure (CPAP) and also in controls of similar visceral adiposity without OSA. Multiple assessments of biomarkers will be made before, during and after sleep. Since it is proposed that the magnitude of these dynamic changes across the sleep period will be affected by degree of visceral obesity and be greater in OSA subjects with cardiovascular comorbidities, studies will be done in 4 groups of subjects: lean and obese with and without such morbidities. In assessing biomarkers the primary outcome variables will be: urinary isoprostanes (oxidative stress); plasma tumor necrosis factor alpha (TNFα) (inflammation); plasma norepinephrine (sympathetic activation); and free fatty acids. Secondary biomarkers will be: Interleukin 6 (IL-6), urinary norepinephrine; urinary normetanephrine; glucose, Intercellular Adhesion Molecule (ICAM), leptin. To complement assessment of circulating biomarkers, an approach utilizing a cellular window will be used. Monocytes will be separated from each blood sample (before, during and after sleep) and RNA extracted. Expression of key genes will be assessed by RT-PCR and microarray studies will be performed in a subset of subjects to assess changes in expression of all genes as a result of OSA. A particular focus will be investigating differences between individuals with OSA with and without cardiovascular comorbidities. Three aspects will be evaluated: a)whether individuals with comorbidities have more oxidative stress and inflammatory change for equivalent degrees of OSA than individuals without such comorbidities; b) whether individuals with comorbidities have lower levels of protective mechanisms-melatonin (an anti-oxidant secreted during sleep), IL-10 (antiinflammatory); c) different gene variants based on a genetic association study using a recently developed CV SNP array. Finally, data will be used to determine whether there is a diagnostic urine and/or blood test for OSA.

ELIGIBILITY:
Inclusion Criteria:

* able to read and write in English
* if female, not pregnant
* goes to bed between 9:30pm-12:30am and sleeps minimum of 7 hours/night
* has telephone access
* BMI < 40

Exclusion Criteria:

* shift worker, irregular schedule
* previous diagnosis of sleep disorder other than OSA
* previous treatment with CPAP, BiPAP, oxygen, surgery for OSA
* current kidney disease, anemia, depression,
* substance abuse/dependence
* BMI > 40
* visual/hearing/cognitive impairments
* smoker who's not willing to refrain from all nicotine during study
* not willing to try CPAP treatment

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OSA patients with moderate to severe disease as confirmed by apnea-hypopnea index (AHI > 15) in a polysomnography. Healthy controls, both snorers and nonsnorers, with an apnea-hypopnea index (AHI < 5) in a polysomnography.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2008-04; Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Magnitude of change in biomarkers during sleep in persons with OSA before & after successful treatment with CPAP, & differences in magnitude of change in persons with different degrees of visceral adiposity, & in those w/ & w/o specific comorbidities. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Allan I Pack, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lim DC, Brady DC, Po P, Chuang LP, Marcondes L, Kim EY, Keenan BT, Guo X, Maislin G, Galante RJ, Pack AI. Simulating obstructive sleep apnea patients' oxygenation characteristics into a mouse model of cyclical intermittent hypoxia. J Appl Physiol (1985). 2015 Mar 1;118(5):544-57. doi: 10.1152/japplphysiol.00629.2014. Epub 2014 Nov 26. PMID 25429097